CLINICAL TRIAL: NCT02413268
Title: Topical Nitroglycerin To Prevent Radial Artery Occlusion After Transradial Access: NTP-RAO Trial
Acronym: NTP-RAO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Total Cardiovascular Solutions (Other)
Responsible Party: Principal Investigator, Dr. Tejas M. Patel, MD, Chairman, Total Cardiovascular Solutions
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NTP1
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Total Atherosclerotic Occlusion of Radial Artery
MeSH Terms: interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Patient receives an antibiotic ointment with no vasoactive drug as a placebo for comparison.
  Interventions: Drug: Nitroglycerin
- Nitropaste (Active Comparator): Nitroglycerin 2% ointment is applied above the compression surface on the skin, to evaluate its efficacy in reducing radial artery occlusion.
  Interventions: Drug: Nitroglycerin

INTERVENTIONS:
Drug: Nitroglycerin
  Other Names: Nitropaste

SUMMARY:
A randomized comparison of topical nitroglycerin versus placebo gel for prevention of radial artery occlusion after transradial catheterization.

DETAILED DESCRIPTION:
Patients and Methods:

Inclusion criteria:

1: All > 18 years old patients referred for transradial coronary angiography.

Exclusion criteria:

1. Absence of informed consent.
2. Known allergy to nitroglycerin.
3. Ad-hoc PCI
4. Previous ipsilateral TRA.
5. Warfarin or NOAC therapy.
6. Systolic blood pressure < 100 mmHg.
7. Critical aortic stenosis (AVA < 0.6 sq.cm)
8. Inability to administer unfractionated heparin.
9. Need for post-procedural use of heparin (UFH, LMWH)
10. Raynaud's disease.
11. Sheathless technique or use of > 11 cm sheath.
12. History of intractable headache of any cause OR Migraine headache.

Transradial Access and Procedure: After routine preparation and sterile draping, the skin of the distal flexor aspect of the forearm was infiltrated with 1-2 ml of preservative free 1% lidocaine, 2-3 fingerbreaths above the styloid process. Radial pulse was palpated at that site and radial artery access was obtained using a 20-gauge teflon sheathed needle after which a 0.021" guide wire was placed through the teflon cannula into the radial artery lumen, once continuous blood flow was visualized. A 5 french, 11 cm hydrophilic introducer sheath (Radiofocus, Terumo Medical) with outer diameter of 2.65 mm will be placed over the guide wire into the radial artery. 2.5 mg of Verapamil and 200 mcg of nitroglycerin were administered via the introducer sheath in an intraarterial fashion. Other equipment will be used as per operator's discretion.

After completion of diagnostic coronary or peripheral angiography, the patients will be randomized to either "Traditional Hemostasis Group" or "Nitropaste Hemostasis Group" using sealed envelope technique (SNOSE). Block randomization will be used for each location.

Hemostasis technique:

Control Group: An inflatable band (TR band, Terumo Medical) will be applied at the radial access site and inflated to obtain hemostasis. Patent hemostasis was attempted in all patients, using the technique described earlier (10). Status of radial artery flow during hemostatic compression will be evaluated at the time of onset of hemostasis, and removal of the band. Duration of compression will be a minimum of 2 hours and upto the operator's discretion.

Nitropaste Group: An inflatable band (TR band, Terumo Medical) will be applied at the radial access site after 0.5 inch aliquot of 2% nitroglycerin ointment is applied uniformly on the surface of the balloon to be in contact with the patients skin. Patent hemostasis will be attempted in all patients, using the technique described earlier (10). Status of radial artery flow during hemostatic compression will be evaluated at the time of onset of hemostasis, and removal of the band. Duration of compression will be a minimum of 2 hours and upto the operator's discretion.

Radial Artery Patency: Radial artery patency after removal of the band and at the time of discharge or 2 hours after removal of the band, whichever comes earlier, will be assessed using reverse Barbeau's test using plethysmographic technique. Ultrasonography will be left upto the operator's discretion.

Primary Study Endpoint:

1: Absence of radial artery antegrade flow as assessed by absence of plethysmographic signal in the index finger after occlusive compression of ipsilateral ulnar artery.

Secondary endpoint:

1. Occurrence of new headache
2. Occurrence of hypotension ( systolic blood pressure < 100 mmHg).

Sample Size Calculation:

Based on the published evidence, 11.3% incidence of RAO at 24 hours after band removal has been observed (Dharma ). Assuming a similar incidence at the time of discharge (< 2 hours after band removal), and a 50% reduction in the primary study endpoint of RAO detected by plethysmography, 1168 patients will need to be randomized, 584 patients in each group, to have a 90% chance of accurately evaluating the difference between the control and treatment arm, using superiority design with an alpha of 5% (10). A cross-over rate of 10% has been used in this calculation. Intent-to-treat and per protocol analyses will be performed, although intent-to-treat analysis will be the primary analysis. Interim analysis will be performed after 600 patients are randomized to assess the safety of either strategy, by a 3 member data monitoring group.

Statistical Analysis Plan:

Data will be expressed in number (percentage) for categorical variables, and as mean ± standard deviation for continuous variables (if normally distributed) or as median ± inter-quartile range (if non-normally distributed). The total study cohort will be categorized into "Control Group" and "NTP Group". Continuous variables will be compared between these 2 groups using student 't' test (if normally distributed) or the Wilcoxon rank-sum test (if non-normally distributed). Categorical variables were compared using chi-squared test or Fischer's exact test as appropriate. Multivariable analyses will be performed to identify predictors of RAO.

ELIGIBILITY:
Inclusion Criteria: Patients referred for cardiac catheterization.

-

Exclusion Criteria:

* 1: Absence of informed consent. 2: Known allergy to nitroglycerin. 3: Ad-hoc PCI 4: Previous ipsilateral TRA. 5: Warfarin or NOAC therapy. 6: Systolic blood pressure < 100 mmHg. 7: Critical aortic stenosis (AVA < 0.6 sq.cm) 8: Inability to administer unfractionated heparin. 9: Need for post-procedural use of heparin (UFH, LMWH) 10: Raynaud's disease. 11: Sheathless technique or use of > 11 cm sheath. 12: History of intractable headache of any cause OR Migraine headache.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Radial Artery Occlusion | up to 2 hours

SECONDARY OUTCOMES:
Headache | up to 4 hours
  Pain in the head that is new-onset
Hypotension | up to 4 hours
  Systolic blood pressure < 90 mmHg that is new-onset

CONTACTS AND LOCATIONS:
Overall Officials: Tejas M Patel, MD, Principal Investigator — Apex Heart Institute, Ahmedabad, India
Locations (1):
- Apex Heart Institute, Ahmedabad, Gujarat, India